CLINICAL TRIAL: NCT03465462
Title: The Influence of Hypotensive Drugs on Zinc, Copper and Iron Status in Experimental and Clinical Studies.
Brief Title: The Influence of Hypotensive Drugs on Mineral Status in Experimental and Clinical Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Collaborators: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Joanna Suliburska, Associate Professor, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 86/09
Record Dates: First submitted 2018-03-01; First posted 2018-03-14 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Nutritional Disorder; Hypertension; Mineral Deficiency
Keywords: hypertension,; zinc; zinc supplementation; antihypertensive monotherapy; mineral status
MeSH Terms: conditions — Nutrition Disorders; Hypertension | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Three stages of the study:
  * stage 1- diagnosis of primary hypertension
  * stage 2 (lasting 3 months) - antihypertensive monotherapy in all subjects
  * stage 3 (lasting 30 days) - 3 groups (3 arms): group/arm C (control group), group/arm D (diet group) and group/arm S (supplementation group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group/arm C (control group) (Active Comparator): Group C in the third stage (30 days) continued drug use with no change in diet and no mineral supplementation.
  Interventions: Dietary Supplement: group/arm C (control group)
- group/arm D (diet group) (Active Comparator): Group D in the third stage (30 days) received an optimal-mineral-content properly balanced diet enriched in food with high zinc content.
  Interventions: Dietary Supplement: group/arm D (diet group)
- group/arm S (supplementation group) (Active Comparator): Group S in the third stage (30 days) received zinc supplementation as one capsule containing 15 mg of Zn taken orally once a day in the morning, two hours after antihypertensive drug administration with no change in diet.
  Interventions: Dietary Supplement: group/arm S (supplementation group)

INTERVENTIONS:
Dietary Supplement: group/arm C (control group) — Group C in the third stage (30 days) continued drug use with no change in diet and no mineral supplementation.
  Arms: group/arm C (control group)
Dietary Supplement: group/arm D (diet group) — Group D in the third stage (30 days) received an optimal-mineral-content properly balanced diet enriched in food with high zinc content.
  Arms: group/arm D (diet group)
Dietary Supplement: group/arm S (supplementation group) — Group S in the third stage (30 days) received zinc supplementation as one capsule containing 15 mg of Zn taken orally once a day in the morning, two hours after antihypertensive drug administration with no change in diet.
  Arms: group/arm S (supplementation group)

SUMMARY:
The aim of the study was to evaluate the effects of hypotensive treatment combined with a higher zinc supply in the diet and supplements on the mineral status and selected biochemical parameters of newly diagnosed hypertensive patients on monotherapy.

DETAILED DESCRIPTION:
The study was designed as a prospective randomized trial and was performed in three stages. In the first stage, primary hypertension was diagnosed and antihypertensive monotherapy was implemented. In the second stage, patients underwent antihypertensive monotherapy lasting three months. The subjects received diuretics; calcium antagonists (Ca-antagonists); angiotensin-converting-enzyme inhibitors (ACE-Is); angiotensin II receptor antagonists (ARBs); or β-blockers. After three months of monotherapy, patients were divided using a randomization list into three equal groups: C (control group), D (diet group) and S (supplementation group). In the third stage, which lasted 30 days, subjects from all groups received the same antihypertensive drug as in the second stage and either an optimal-mineral-content diet (group D), zinc supplementation (group S), or continued drug use with no change in diet and no mineral supplementation (group C). Patients from group D received an optimal-mineral-content properly balanced diet enriched in food with high zinc content prepared individually for each patient by a qualified dietician. Patients from group S received zinc supplementation as one capsule containing 15 mg of Zn taken orally once a day in the morning, two hours after antihypertensive drug administration with no change in diet, through all 30 days of the third stage of the trial.

During the study, patients were asked to not use dietary supplements and not to change their lifestyle or level of physical activity. On the last day of each stage of the study, blood, urine, and hair samples were collected from the subjects, and blood pressure and anthropometric parameters were measured.

ELIGIBILITY:
Inclusion Criteria:

* informed written consent;
* age 18-65 years;
* primary hypertension;
* beginning monotherapy with an antihypertensive drug;
* stable body weight (less than 3 kg self-reported change during the three months prior to enrollment).

Exclusion Criteria:

* any secondary form of hypertension;
* the use of mineral supplements within the three months prior to enrollment;
* lipid disorders requiring treatment in the three months prior to the trial;
* a history of ischemic heart disease, stroke, congestive heart failure,
* clinically significant arrhythmia or conduction disorders, peripheral artery or vein disease, diabetes mellitus, abnormal renal, liver or thyroid gland function,
* clinically significant chronic or acute inflammatory process within the respiratory, genitourinary, or digestive tract, or in the oral cavity, larynx, pharynx, or in the paranasal sinuses, or connective tissue diseases, arthritis, or malignancy;
* infection in the month prior to enrollment,
* having an pacemaker implanted;
* alcohol, nicotine or drug abuse;
* mental disorders;
* pregnancy, childbirth or lactation at enrollment or in the three months prior to enrollment;
* or any other condition that, in the opinion of investigators, would make participation in the study not in the best interest of the subject, or could prevent, limit, or confound the efficacy of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Serum zinc- stage I | At baseline
  Serum zinc concentration in stage I of the trial
Serum zinc- stage II | After 3 months
  Serum zinc concentration in stage II of the trial
Serum zinc- stage III | After 3 months and 30 days
  Serum zinc concentration in stage III of the trial

SECONDARY OUTCOMES:
Body mass- stage I | At baseline
  Body mass in stage I
Body mass- stage II | After 3 months
  Body mass in stage II
Body mass- stage III | After 3 months and 30 days
  Body mass in stage III
Body height- stage I | At baseline
  Body height in stage I
Body height- stage II | After 3 months
  Body height in stage II
Body height- stage III | After 3 months and 30 days
  Body height in stage III
Blood pressure- stage I | At baseline
  Blood pressure in stage I
Blood pressure- stage II | After 3 months
  Blood pressure in stage II
Blood pressure- stage III | After 3 months and 30 days
  Blood pressure in stage III
Erythrocytes zinc- stage I | At baseline
  Zinc concentration in erythrocytes in stage I
Erythrocytes zinc- stage II | After 3 months
  Zinc concentration in erythrocytes in stage II
Erythrocytes zinc- stage III | After 3 months and 30 days
  Zinc concentration in erythrocytes in stage III
Urine zinc- stage I | At baseline
  Zinc concentration in urine in stage I
Urine zinc- stage II | After 3 months
  Zinc concentration in urine in stage II
Urine zinc- stage III | After 3 months and 30 days
  Zinc concentration in urine in stage III
Hair zinc- stage I | At baseline
  Zinc content in hair in stage I
Hair zinc- stage II | After 3 months
  Zinc content in hair in stage II
Hair zinc- stage III | After 3 months and 30 days
  Zinc content in hair in stage III
Serum iron- stage I | At baseline
  Iron concentration in serum in stage I
Serum iron- stage II | After 3 months
  Iron concentration in serum in stage II
Serum iron- stage III | After 3 months and 30 days
  Iron concentration in serum in stage III
Erythrocytes iron- stage I | At baseline
  Iron concentration in erythrocytes in stage I
Erythrocytes iron- stage II | After 3 months
  Iron concentration in erythrocytes in stage II
Erythrocytes iron- stage III | After 3 months and 30 days
  Iron concentration in erythrocytes in stage III
Urine iron- stage I | At baseline
  Iron concentration in urine in stage I
Urine iron- stage II | After 3 months
  Iron concentration in urine in stage II
Urine iron- stage III | After 3 months and 30 days
  Iron concentration in urine in stage III
Hair iron- stage I | At baseline
  Iron content in hair in stage I
Hair iron- stage II | After 3 months
  Iron content in hair in stage II
Hair iron- stage III | After 3 months and 30 days
  Iron content in hair in stage III
Serum copper- stage I | At baseline
  Serum copper concentration in stage I
Serum copper- stage II | After 3 months
  Serum copper concentration in stage II
Serum copper- stage III | After 3 months and 30 days
  Serum copper concentration in stage III
Erythrocytes copper- stage I | At baseline
  Erythrocytes copper concentration in stage I
Erythrocytes copper- stage II | After 3 months
  Erythrocytes copper concentration in stage II
Erythrocytes copper- stage III | After 3 months and 30 days
  Erythrocytes copper concentration in stage III
Urine copper- stage I | At baseline
  Urine copper concentration in stage I
Urine copper- stage II | After 3 months
  Urine copper concentration in stage II
Urine copper- stage III | After 3 months and 30 days
  Urine copper concentration in stage III
Hair copper- stage I | At baseline
  Hair copper content in stage I
Hair copper- stage II | After 3 months
  Hair copper content in stage II
Hair copper- stage III | After 3 months and 30 days
  Hair copper content in stage III
Glucose- stage I | At baseline
  Glucose serum concentration in stage I
Glucose- stage II | After 3 months
  Glucose serum concentration in stage II
Glucose- stage III | After 3 months and 30 days
  Glucose serum concentration in stage III
C-reactive protein- stage I | At baseline
  C-reactive protein serum concentration in stage I
C-reactive protein- stage II | After 3 months
  C-reactive protein serum concentration in stage II
C-reactive protein- stage III | After 3 months and 30 days
  C-reactive protein serum concentration in stage III

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Suliburska, Assoc. Prof., Study Chair — Poznan University of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland